CLINICAL TRIAL: NCT04238741
Title: Audio-recording of Consent for Anaesthesia for Elective Caesarean Section - a Pilot Study
Brief Title: Audio-recording of Consent for Anaesthesia for Elective Caesarean Section
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chelsea and Westminster NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C&W18/033
Record Dates: First submitted 2018-11-06; First posted 2020-01-23 (Actual); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Caesarean Section; Anesthesia
MeSH Terms: interventions — Anesthesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Audio-recording of consent for anaesthesia for elective caesarean section — Antenatal women will be invited to attend 5-15 days before their caesarean section for an anaesthetic consent discussion with audio-recording. Participants will complete a questionnaire immediately following the recorded discussion and again within the 48 hours following their surgery, to establish their views on the process of audio-recording of consent and the potential usefulness/acceptability of the audio-recording.

SUMMARY:
Informed consent should be obtained from patients (with capacity) before treatment - including anaesthesia - is administered. If the consent process is inadequate, it may lead to poor decision-making and dissatisfaction, sometimes leading to complaints or legal claims. Obstetric practice is a high-risk area for medicolegal claims and accurate, reliable documentation of consent is therefore vital in this group.

The hypothesis is that audio-recording of consent discussions would provide a record of the discussion for the patient and healthcare staff to refer to later, to assist in understanding and potentially prevent dissatisfaction, complaints and claims; and may improve the consent process itself if both parties know that the discussion will be audio-recorded.

This project aims to establish the acceptability and feasibility of audio-recording of consent for elective caesarean section. The investigators will trial the concept by establishing audio-recording of consent for anaesthesia for elective caesarean section, and aim to investigate the views of patients at Chelsea and Westminster Hospital taking part.

The investigators aim to address the following research questions:

* what are the views of patients (and to a lesser extent, doctors) involved in audio-recording of consent discussions for anaesthesia for elective caesarean section regarding its acceptability and utility?
* what were the perceived concerns and/or practical obstacles to overcome in the trial of concept?

DETAILED DESCRIPTION:
This is a pilot study to trial audio-recording of consent and evaluate its potential for use in day to day clinical care. This study will be a quantitative, observational survey of 20 antenatal maternity patients scheduled for elective caesarean section, who have attended 5-15 days before their planned surgery for anaesthetic consent discussions with audio-recording. Participants will complete a questionnaire immediately following the recorded discussion and again within the 48 hours following surgery. The study aims to establish participants' views on the process of audio-recording of consent and the potential usefulness/acceptability of the audio-recording.

The antenatal maternity patients will be a random/convenience sample of women booked for elective caesarean section at Chelsea and Westminster Hospital. These women will be expected to have a fairly uniform consent discussion with an anaesthetist before their surgery. Participants will be selected according to the date of the planned caesarean section, their availability and that of the research team, in turn until 20 women have completed the study (i.e. have had a recorded discussion, undergone elective caesarean section, and completed the postnatal questionnaire).

The doctors involved in consent discussions will be a small group of anaesthetists (n = 3) to maintain consistency; these anaesthetists will also complete questionnaires in order to raise any themes/issues for further evaluation, whilst accepting that the sample size will be too small for firm conclusions.

The questionnaires will be completely anonymous and have been designed to minimise bias in the question wording and structure, with input from patients and staff in the design process. An anaesthetist will be on hand to facilitate completion of the questionnaires and to assist with understanding of the questions.

ELIGIBILITY:
Inclusion Criteria:

* maternity patients: antenatal patients before elective caesarean section (5-15 days)
* doctors: anaesthetists who cover labour ward

Exclusion Criteria:

* maternity patients not planning caesarean section
* those booked for elective caesarean section less than a week in advance of the date
* those who do not have the facility to listen to a CD
* those with limited understanding of English
* any woman with a hearing impairment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 29 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-01-29 (Actual); Study Completion 2019-01-29 (Actual)

PRIMARY OUTCOMES:
Views of patients regarding the acceptability and utility of audio-recording of consent discussions for anaesthesia for elective caesarean section. | Up to 6 months
  Participants' views on the acceptability and utility of audio-recording of consent discussion for anaesthesia for elective caesarean section will be established using questionnaires completed immediately after the recorded discussion and again within the 48 hours following their caesarean section. The questions will include numeric rating scales, with participants required to indicate how strongly they agree/disagree with, and how positively/negatively they feel about a number of statements (where 1 = strongly agree/very positive and 10 = strongly disagree/very negative).

SECONDARY OUTCOMES:
Views of doctors regarding the acceptability and utility of audio-recording of consent discussions for anaesthesia for elective caesarean section. | Up to 6 months
  The views of doctors involved in audio-recording of consent discussions will be sought on completion of the trial using a questionnaire.The questions will include numeric rating scales, with participants required to indicate how strongly they agree/disagree with, and how positively/negatively they feel about a number of statements (where 1 = strongly agree/very positive and 10 = strongly disagree/very negative).
Perceived concerns and/or practical obstacles to overcome in the trial of concept | Up to 6 months
  Questionnaires given to patients and doctors involved in the trial will ask specifically about any concerns and practical obstacles that they feel need to be overcome.The questions will include numeric rating scales, with participants required to indicate how strongly they agree/disagree with, and how positively/negatively they feel about a number of statements (where 1 = strongly agree/very positive and 10 = strongly disagree/very negative).

CONTACTS AND LOCATIONS:
Overall Officials: Steve Yentis, Principal Investigator — Chelsea and Westminster Hospital
Locations (1):
- Chelsea and Westminster Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No